CLINICAL TRIAL: NCT00460421
Title: A Phase 1 Dose-escalation Study to Evaluate the Safety and Pharmacokinetics (PK) of Palifermin in Pediatric Subjects With Acute Leukemias Undergoing Myeloablative Therapy and Allogeneic Hematopoietic Stem Cell Transplant (HSCT)
Brief Title: A Phase 1 Dose-escalation Study to Evaluate the Safety and Pharmacokinetics (PK) of Palifermin in Subjects With Acute Leukemias Undergoing HSCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20010133; NCT00896506 (obsolete NCT alias)
Record Dates: First submitted 2007-04-12; First posted 2007-04-16 (Estimated); Results first posted 2012-07-03 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-11

CONDITIONS: Leukemia
Keywords: Oral Mucositis; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Palifermin; Kepivance
MeSH Terms: conditions — Leukemia; Stomatitis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Fibroblast Growth Factor 7; Whole-Body Irradiation; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Palifermin Dose Escalation (Experimental): A 3 dose escalation design. Sucessive cohorts of patient (9 patients per group) will each be administered Palifermin as an IV bolus injection (40, 60 or 80 µg) once daily for 3 consecutive days before the start of conditioning regimen (chemotherapy and total body irradiation) and after HCST (Day -10, -9, -8 and Day 0, +1, +2 respectively).
  Interventions: Drug: Palifermin; Radiation: Total Body irradiation; Drug: Chemotherapy

INTERVENTIONS:
Drug: Palifermin — Palifermin will be administered as an IV bolus injection (40, 60 or 80 µg/kg/day)once daily for 3 consecutive days before the start of conditioning regimen and after HCST (Day -10, -9, -8 and Day 0, +1, +2 respectively).
  Other Names: Kepivance
Radiation: Total Body irradiation
Drug: Chemotherapy — High dose etoposide, Cyclophosphamide

SUMMARY:
20010133 is an open-label, dose escalation study in pediatric patients with acute leukemias receiving myelotoxic therapy (high dose etoposide, cyclophosphamide and total body irradiation [TBI]) followed by hematopoietic stem cell transplant (HSCT). The study will evaluate the safety and pharmacokinetics of palifermin in pediatric patients. Three doses (40 μg/kg/day, 60 μg/kg/day, and 80 μg/kg/day) are to be evaluated in each age group (1 to 2, 3 to 11, and 12 to 16 years, respectively) using a conventional dose escalation design. Palifermin is administered for 3 consecutive days (Day -10 to Day -8, respectively) before the start of the conditioning regimen and for 3 consecutive days (Day 0 to Day +2) following HSCT. Patients will be enrolled simultaneously to each age group to identify a safe, well tolerated, efficacious dose in each age group. Patients will also be followed for secondary malignancies, progression-free survival (PFS) and overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

1. Acute lymphoblastic leukemia (ALL) or acute myeloid leukemia (AML) requiring HSCT
2. Age ≥ 1 and ≤ 16 years at screening
3. Lansky performance status > 60%
4. Candidate for allogeneic HSCT protocol:

   * Adequate kidney function: Serum creatinine: ≤ 1.5 mg/dL or creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 60 mL/min/1.73m2
   * Adequate liver function: Serum total bilirubin: ≤ 2.0 mg/dl; aspartate transaminase (AST)/alanine aminotransferase (ALT) ≤ 4.0 x institutional upper limits of normal (IULN); Albumin ≥ 2 g/dL
   * Adequate cardiac function: shortening fraction > 29% documented by echocardiogram, or ejection fraction ≥ 50% documented by multigated acquisition scan (MUGA).
   * Adequate pulmonary function documented by corrected lung diffusion capacity test (DLCO) > 50% or oxygen saturation of ≥ 92% on room air if unable to perform pulmonary function tests
   * Negative for human immunodeficiency virus (HIV), hepatitis C virus (HCV), human T cell lymphotropic virus (HTLV)
5. Identification of an HLA-compatible donor per institutional standards
6. Assent from a minor (if the child is capable of giving assent) per Department of Health and Human Services (DHHS) guidelines listed in 21CFR 50.55 and local Institutional Review Board (IRB) standards.
7. Serum amylase and lipase: ≤ 1.2 x IULN
8. Negative serum/urine pregnancy test for females with childbearing potential within 4 days before administration of the first palifermin dose
9. Agreement by males and females of reproductive potential to use an effective means of contraception 30 days prior to enrollment through Day +30 (end of treatment)

Exclusion Criteria:

1. Prior treatment with palifermin or other keratinocyte growth factors
2. Received an investigational product or device, with the exception investigational stem cell separators, in another clinical trial within 30 days before enrollment.
3. Known to have a life threatening infection not responding well to treatment
4. Past history of veno-occlusive disease of the liver
5. Known sensitivity to any Escherichia coli-derived products with grade 3 to 4 allergies to L-asparaginase [grade 1 to 2 allergies to L-asparaginase will be allowed].
6. Receiving glutamine or any other medication to reduce the incidence of oral mucositis (OM) within 30 days before enrollment
7. Previous or concurrent malignancy other than entry diagnostic criteria and/or solid organ transplantation and/or treatment of congenital immunodeficiency
8. History of pancreatitis
9. Breastfeeding (giving)

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2006-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maarten de Chateau, MD, PhD, Study Director — Swedish Orphan Biovitrum AB
Locations (7):
- United States (7):
  - Arizona Cancer Center, Tucson, Arizona
  - Loma Linda University, Loma Linda, California
  - Children´s Hospital, Los Angeles, California
  - Regents of University of California, Los Angeles, California
  - Children´s Hospital of Orange, Orange, California
  - Children´s Memorial, Chicago, Illinois
  - University of Texas, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase 1 dose-escalation study to evaluate the safety and pharmacokinetics (PK) of palifermin in pediatric subjects with acute leukemias undergoing myeloblative therapy and allogeneic hematopoietic stem cell transplant (HSCT) was performed in 7 centers in USA between 2006 and 2011.
Groups:
- Palifermin 40 µg/kg/Day; Palifermin 60 µg/kg/Day; Palifermin 80 µg/kg/Day: Three subjects from each age group (1-2, 3-11, 12-16 years) were sequentially enrolled into the 3 planned dosing cohorts
Period: Overall Study
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day
Started | 9 | 9 | 9
Completed | 9 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day | Total
Number analyzed (Participants) | 9 | 9 | 9 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 9 | 27
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.4 (6.3) | 7.4 (5.6) | 8.0 (6.6) | 7.6 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 12
  Male | 6 | 5 | 4 | 15
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose Limiting Toxicities (DLTs)
Description: A DLT is appearance of side effects during treatment severe enough to prevent further increase in dosage or strength of treatment agent, or to prevent continuation of treatment at any dosage level.
  A DLT was defined as: Grade 3 or 4 AE [based on Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (CTCAE) v3.0] considered by the investigator to be related to palifermin with the exceptions: Grade 3 erythema, pruritus or rash that resolves within 7 days of the last dose of palifermin.
  The percentage of particiapnts with a DLT during the study was assessed.
Time Frame: Approximately 1 month duration (Day -10 through Day +16)
Population: Safety Analysis Set. This set consisted of subjects who received at least one dose of palifermin.
Measure: Number; unit: percentage of participants
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day
Number analyzed (Participants) | 9 | 9 | 9
percentage of participants | 0 | 0 | 0

2. Secondary Outcome: Incidence of Serum Palifermin Antibody Formation
Description: The percentage of participants developing palifermin antibodies during the study was assessed.
Time Frame: Approximately 4 month duration (Through Day + 100 (+/- 40 days))
Population: Safety Analysis Set. This set consisted of subjects who received at least one dose of palifermin.
Measure: Number; unit: percentage of participants
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day
Number analyzed (Participants) | 9 | 9 | 9
percentage of participants | 0 | 0 | 0

3. Secondary Outcome: Incidence of Severe Adverse Events (AEs)
Description: The percentage of participants with a severe AE during the study was assessed.
Time Frame: Approximately 1 1/2 months duration (Through Day +30/End of Treatment)
Population: Safety Analysis Set. This set consisted of subjects who received at least one dose of palifermin.
Measure: Number; unit: percentage of participants
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day
Number analyzed (Participants) | 9 | 9 | 9
percentage of participants | 100 | 100 | 100

4. Secondary Outcome: Incidence of Laboratory Abnormalities
Description: The percentage of participants with a laboratory value outside the normal ranges during the study.
Time Frame: Approximately 1 1/2 months duration (Through Day +30/End of Treatment)
Population: Safety Analysis Set. This set consisted of subjects who received at least one dose of palifermin.
Measure: Number; unit: percentage of participants
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day
Number analyzed (Participants) | 9 | 9 | 9
percentage of participants | 100 | 100 | 100

5. Secondary Outcome: Pharmacokinetics of Palifermin, Clearence (CL) After the 1st Intravenous (IV) Bolus Injection for Multiple Dose Levels
Description: Clearence was estimated as dose divided by the area under serum concentration-time curve from time zero to infinity where the dose was given in amount palifermin actually administered.
Time Frame: Day -10
Population: Pharmacokinetic Analysis Set. This set consists of all subjects who receive at least one dose of palifermin and who have a sufficient number of serum concentration data points to allow calculation of the pharmacokinetic variables.
Measure: Median (Full Range); unit: mL/hr/kg
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day
Number analyzed (Participants) | 9 | 9 | 9
mL/hr/kg | 1954.84 [570.83 to 3629.06] | 2164.87 [419.39 to 5152.07] | 3932.30 [1268.22 to 18182.41]

6. Secondary Outcome: Pharmacokinetics of Palifermin, Volume of Distribution at Steady State (Vss) After the 1st IV Bolus Injection for Multiple Dose Levels
Time Frame: Day -10
Population: as for outcome 5
Measure: Median (Full Range); unit: mL/kg
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day
Number analyzed (Participants) | 9 | 9 | 9
mL/kg | 2552.79 [369.31 to 4862.29] | 5134.84 [1033.25 to 28349.41] | 8580.91 [1165.08 to 70085.13]

7. Secondary Outcome: Pharmacokinetics of Palifermin, Terminal Half-life (t½,z) After the 1st IV Bolus Injection for Multiple Dose Levels
Description: The terminal half-life was calculated as ln(2)/lambda,z where lambda,z was estimated using at least three quantifiable serum concentrations of the terminal log-linear phase.
Time Frame: Day -10
Population: as for outcome 5
Measure: Median (Full Range); unit: hour
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day
Number analyzed (Participants) | 9 | 9 | 9
hour | 2.91 [1.43 to 5.81] | 3.05 [2.19 to 8.36] | 3.68 [0.97 to 4.88]

8. Secondary Outcome: Pharmacokinetics of Palifermin, t½,z After the 3rd IV Bolus Injection for Multiple Dose Levels
Description: as for outcome 7
Time Frame: Day -8
Population: as for outcome 5
Measure: Median (Full Range); unit: hour
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day
Number analyzed (Participants) | 9 | 9 | 9
hour | 3.40 [0.84 to 5.71] | 3.89 [3.21 to 11.84] | 2.99 [2.06 to 4.03]

9. Secondary Outcome: Pharmacokinetics of Palifermin, Area Under the Concentration Time Curve From Zero to the End of the Dosing Interval (AUCtau) After the 1st IV Bolus Injection for Multiple Dose Levels
Description: The AUC was estimated using the linear/log trapezoidal method for AUC0-tau from time zero to the end of the dosing interval (24 hours (hrs) post-dose)
  Data collected at time points: 0, 2 minutes (min), 15 min, 30 min, 60 min, 2 hrs, 4 hrs, 6, hrs, 10, hrs and 24 hrs post-dose.
Time Frame: Day -10
Population: as for outcome 5
Measure: Median (Full Range); unit: ng*hr/mL
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day
Number analyzed (Participants) | 9 | 9 | 9
ng*hr/mL | 16.54 [4.69 to 70.57] | 18.14 [12.35 to 142.71] | 38.44 [4.53 to 185.35]

10. Secondary Outcome: Pharmacokinetics of Palifermin, AUCtau After the 3rd IV Bolus Injection for Multiple Dose Levels
Description: as for outcome 9
Time Frame: Day -8
Population: as for outcome 5
Measure: Median (Full Range); unit: ng*hr/mL
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day
Number analyzed (Participants) | 9 | 9 | 9
ng*hr/mL | 18.32 [1.73 to 63.65] | 17.97 [2.45 to 325.96] | 34.74 [3.14 to 295.11]

11. Secondary Outcome: Long-Term Follow-Up: Incidence of Secondary Malignancies
Time Frame: Up to 4 years duration (Assessments performed on months 6, 9, 12 (+/- 30 Days) for the first year and then annually)
Population: Safety Analysis Set. This set consisted of subjects who received at least one dose of palifermin.
Measure: Number; unit: percentage of participants
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day
Number analyzed (Participants) | 9 | 9 | 9
percentage of participants | 0 | 11 | 0

12. Secondary Outcome: Long-Term Follow-Up: Progression Free Survival
Description: Progression free survival (PFS) was defined as the number of days between the date of first investigational product administration and the date when physical or radiological evidence of disease progression is determined or death (regardless of cause)
Time Frame: Up to 4 years duration (Assessments performed on months 6, 9, 12 (+/- 30 Days) for the first year and then annually)
Population: Safety Analysis Set. This set consisted of subjects who received at least one dose of palifermin.
Measure: Median (Full Range); unit: months
Groups:
- All Subjects: All subjects from each age group (1-2, 3-11, 12-16 years)
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day | All Subjects
Number analyzed (Participants) | 9 | 9 | 9 | 27
months | NA [NA to NA] — Reported for the entire study population | NA [NA to NA] — Reported for the entire study population | NA [NA to NA] — Reported for the entire study population | 36 [6 to 48]

13. Secondary Outcome: Long-Term Follow-Up: Overall Survival
Description: Overall survival was defined as the number of days from the date of first investigational product administration to the date of death (regardless of cause)
Time Frame: Up to 4 years duration (Assessments performed on months 6, 9, 12 (+/- 30 Days) for the first year and then annually)
Population: Safety Analysis Set. This set consisted of subjects who received at least one dose of palifermin.
Measure: Median (Full Range); unit: months
Arm/Group | Palifermin 40 µg/kg/Day | Palifermin 60 µg/kg/Day | Palifermin 80 µg/kg/Day | All Subjects
Number analyzed (Participants) | 9 | 9 | 9 | 27
months | NA [NA to NA] — Reported for the entire study population | NA [NA to NA] — Reported for the entire study population | NA [NA to NA] — Reported for the entire study population | 36 [6 to 48]

ADVERSE EVENTS:
Time Frame: Adverse events collected from signed informed consent to Day 30, i.e. a period of up to 71 days.
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 5/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=27)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Enterococcal infection (Infections and infestations) | 1 (1)
Septic chock (Infections and infestations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Venoocclusive disease (Vascular disorders) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=27)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Pericardial effusion (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 7
Ear pain (Ear and labyrinth disorders) | 2
Dry eye (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 15
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 19
Dyspepsia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Gingival hyperplasia (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 2
Lip dry (Gastrointestinal disorders) | 2
Mouth haemorrhage (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 21
Oesophagitis (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 2
Perianal erythema (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 23
Catheter related complication (General disorders) | 6
Catheter site pain (General disorders) | 5
Chills (General disorders) | 3
Face oedema (General disorders) | 3
Fatigue (General disorders) | 7
Irritability (General disorders) | 4
Oedema (General disorders) | 4
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 4
Pyrexia (General disorders) | 22
Hepatomegaly (Hepatobiliary disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 5
Acute graft versus host disease in skin (Immune system disorders) | 5
Alpha haemolytic streptococcal infection (Infections and infestations) | 3
Bacteraemia (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 3
Enterococcal sepsis (Infections and infestations) | 3
Fungal infection (Infections and infestations) | 2
Parotitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 3
Staphylococcal infection (Infections and infestations) | 4
Urinary tract infection enterococcal (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 4
Head injury (Injury, poisoning and procedural complications) | 2
Blood bilirubin increased (Investigations) | 2
Occult blood positive (Investigations) | 2
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 18
Decreased appetite (Metabolism and nutrition disorders) | 2
Fluid retention (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 10
Hyponatraemia (Metabolism and nutrition disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
bone pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 11
Lethargy (Nervous system disorders) | 2
Agitation (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 4
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 3
Renal tubular acidosis (Renal and urinary disorders) | 2
Scrotal erythema (Reproductive system and breast disorders) | 2
Testicular pain (Reproductive system and breast disorders) | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 4
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 3
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2
Petechiae (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 16
Rash (Skin and subcutaneous tissue disorders) | 15
Skin disorder (Skin and subcutaneous tissue disorders) | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 16
Hypotension (Vascular disorders) | 7

LIMITATIONS AND CAVEATS:
The original protocol included a long term follow-up (LTFU) phase up to 10 years. This was reduced in a protocol amendment to up to the time when the last enrolled subject had completed the day +100 follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits sponsor a limited period of time to review material discussing trial results (approximately up to 90 days). Sponsor may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, investigator agrees not to publish any results before the first multi-center publication.